CLINICAL TRIAL: NCT06085846
Title: Real-World Registry - The Vivally® System
Status: Enrolling by invitation | Type: Observational
Sponsor: Avation Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AMOAB2301
Record Dates: First submitted 2023-10-04; First posted 2023-10-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Urinary Incontinence; Urinary Urge Incontinence
Keywords: Neuromodulation; Overactive Bladder; Overactive Bladder Syndrome; Wearable; Non-invasive; Mobile Application; Electronic Bladder Diary; Urgency
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Vivally® System Wearable, Non-Invasive Neuromodulation System, and Mobile Application — Vivally® System Wearable, Non-Invasive Neuromodulation System and Mobile Application to treat patients with the conditions of urinary incontinence and urinary urgency.

SUMMARY:
This is a Real-World Registry Study to collect real-world dosing, utilization, demographic, quality of life, and data from the e-bladder diaries of patients utilizing the Vivally® System. Data points will be drawn from the Avation Medical HIPAA-compliant cloud database including but not limited to:

Therapy compliance and stimulation metrics

Diary entries provided by patients

Various questionnaires

Participants have the option to opt out of allowing their data to be part of any publication at any time.

DETAILED DESCRIPTION:
Collect real-world dosing, utilization, demographics and quality of life data from the eDiaries of patients utilizing the Vivally® System.

Gather feedback from patients on their experience and satisfaction with the Vivally® System therapy

Identify trends in dosing, compliance, and therapy parameters in order to optimize the wearable, Vivally® System neuromodulation therapy for participants

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the Real-World Registry Study, Participants must satisfy all of the following criteria:

* Are an appropriate candidate for the Vivally® System as determined, and prescribed by a licensed clinical professional
* Have provided informed consent to have their data included in publications associated with this study

Exclusion Criteria:

While it is up to the discretion of the clinician to prescribe the Vivally® System for a specific patient, the Vivally® System is contraindicated for use on patients who have the following history or conditions:

* Patients with pacemakers of implanted defibrillators
* Patients with nerve damage that could impact either transcutaneous tibial nerve stimulation or pelvic floor function
* This product is not intended for intra-cardiac or trans-thoracic use

Additional contraindications, warnings and precautions are listed in the User Guide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person that has been prescribed the Vivally® System by a licensed clinical professional and who provides Informed Consent to allow collection of various data points for future publication.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2043-07-01 (Estimated); Study Completion 2043-07-01 (Estimated)

PRIMARY OUTCOMES:
Real-world Usage | Length of Study, on average 20 years
  Collect real-world dosing, utilization, demographics and quality of life data from the eDiaries of patients utilizing the Vivally® System.

SECONDARY OUTCOMES:
Patient Satisfaction | Length of Study, on average 20 years
  Gather feedback from patients on their experience and satisfaction with the Vivally® System therapy.
Prescribing Trends | Length of Study, on average 20 years
  Identify trends in dosing in order to optimize the wearable, Vivally® System neuromodulation therapy for prescribers. Dosing consists of therapy pulse width parameters (μs) and therapy schedule (sessions completed per week).
Patient Compliance | Length of Study, on average 20 years
  Identify trends in patient compliance in order to optimize the wearable, Vivally® System neuromodulation therapy for participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Avation Medical, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No